CLINICAL TRIAL: NCT05657184
Title: An Open-label Clinical Study to Explore the Safety, Tolerability and Preliminary Efficacy of REGEND001 for Treatment of Idiopathic Pulmonary Fibrosis (IPF).
Brief Title: Treatment of Idiopathic Pulmonary Fibrosis (IPF) by REGEND001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regend Therapeutics (Industry)
Collaborators: Peking Union Medical College Hospital (Other); Ruijin Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Regend Therapeutics XLotus (Jiangxi) Co, Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XHYX-IND-IPF-P1
Record Dates: First submitted 2022-11-15; First posted 2022-12-20 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- REGEND001 (Experimental): Transplantation of autologous airway basal cells
  Interventions: Drug: REGEND001

INTERVENTIONS:
Drug: REGEND001 — Transplantation of REGEND001 for dose escalation.

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a condition where the lungs are damaged and scarred with unknown reason, making breathing becomes increasingly difficult.. REGEND001, made from airway basal cells with ability to regenerate lung tissue, is promising to IPF treatment. In this study, a single-armed clinical trial is ongoing to assess the safety and tolerability of REGEND001 in treatment of IPF. Different doses of REGEND001 is evaluated to establish a dose-response relationship and to suggest appropriate dose for subsequent clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged between 50 to 75.
* Diagnosis of IPF according to 2018 Idiopathic Pulmonary Fibrosis Diagnostic Guidelines.
* Participants with 30%~79% of the predicted value in diffusing capacity for carbon monoxide (DLCO) and more than 50% of the predicted value in forced vital capacity (FVC) in pulmonary function tests within 3 months before screening.
* Participants with typical HRCT images of IPF in the past 12 months.
* Participants tolerant to bronchofiberscopy.
* Participants fully informed with the purpose, method and possible discomfort of the trial, agreeing to participate in the trial and signing the informed consent voluntarily.
* Participants with good adherence, willing to take medication and regular follow-up examinations as required by the protocol.
* Participants able to understand and cooperate with the completion of pulmonary function tests.

Exclusion Criteria:

* Participants who cannot tolerate cell therapy.
* Pregnant or lactating women.
* Participants with syphilis or any of human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV) positive antibody; of which stable HBV carriers after drug treatment and cured hepatitis C patients can be enrolled.
* Participants with malignant tumors or a history of malignant tumors.
* Participants with a history of long-term use of drugs known to cause pulmonary fibrosis, such as amiodarone before screening.
* Participants with lung infections or other infections, including bacterial and viral infections, with requirement of intravenous medications before cell transplantation.
* Participants with a history of invasive or noninvasive mechanical ventilation within 4 weeks.
* Participants with any of the following lung diseases: asthma, active tuberculosis, pulmonary embolism, pneumothorax, pulmonary hypertension, pneumoconiosis, etc.; lung cancer, bronchiolitis obliterans or other active lung disease; pneumonia currently or in the past 4 weeks; pneumonectomy previously.
* Requirement of oxygen therapy for more than 15 hours per day.
* Suffering from serious diseases of other system.
* leukopenia or agranulocytosis of any cause; blood creatinine > 2.5 times the upper limit of normal; alanine transaminase (ALT) and aspartate transaminase (AST) > 2.5 times the upper limit of normal in the laboratory tests.
* Participants with a history of mental illness, suicide risk, epilepsy or other central nervous system disorders.
* Severe arrhythmias (such as ventricular tachycardia, frequent supraventricular tachycardia, atrial fibrillation, atrial flutter, etc.) or atrioventricular block of degree II or above, shown by 12-lead Electrocardiogram (ECG).
* Participants with a history of abusing alcohol or illicit drug.
* Participants allergic to cattle products.
* Participants in other clinical trials in the past 3 months.
* Participants with poor compliance and difficult to complete the trial.
* Investigators, employees of research centers or family members of them (none of whom are suitable to participate in the trial to ensure the objectivity of the research);
* Participants with a history of hospitalization owing to acute exacerbation of IPF or other respiratory diseases three or more times within the past year.
* Participants who is taking or is goning to take nintedanib within a month.
* Participants with other acquired or congenital immunodeficiency disorders, or with a history of organ transplantation or cell transplantation therapy.
* Participants whose expected survival may be less than one year judged by the investigator.
* Male participants of childbearing potential and female participants within childbearing age were reluctant to use effective contraception from the time of signing the informed consent to 6 months after cell therapy.
* Participants assessed to be inappropriate in this clinical trial by investigator.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of the cell therapy-related adverse events (AEs) | Within 24 weeks after treatment
  Dose escalation is based on incidence of cell therapy-related AEs. Severity of cell therapy-related adverse events (AEs) is evaluated according to Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
Incidence of complication related to bronchoscopy | Within 24 weeks after treatment
  REGEND001 is given to subjects by bronchoscopy. Thus, incidence of complication related to bronchoscopy is adapted to assess the safety of the products.
Change in lung diffusing capacity for single-breath carbon monoxide (DLCO-sb) from baseline | 4, 12 and 24 weeks after treatment
  DLCO-sb is measured by the single-breath method. It is considered a measure of the conductance of CO across the alveolar-capillary membrane and its binding with hemoglobin.
Change in forced vital capacity (FVC) from baseline | 4, 12 and 24 weeks after treatment
  FVC indicates the volume of air that can forcibly be blown out after a full inspiration.
Change in the ratio of diffusing capacity for carbon monoxide/ the alveolar volume (DLCO/VA) from baseline | 4, 12 and 24 weeks after treatment
  The DLCO test refers to the diffusing capacity for carbon monoxide in the lungs. It is a type of pulmonary function test that helps to assess how well gas is exchanged between the lungs and the bloodstream. Since DLCO is affected by the amount of inhaled gas and lung volume, the alveolar ventilation is considered to exclude the effect of lung volume on diffusion volume in evaluating diffusion function.
Change in 6-minute-walk test (6MWT) from baseline | 4, 12 and 24 weeks after treatment
  The 6MWT is a commonly used test for the objective assessment of functional exercise capacity by testing the distance patients can walk at the fastest speed within 6 minutes.
Change in St. George's Respiratory Questionnaire (SGRQ) scale from baseline | 4, 12 and 24 weeks after treatment
  Quality of life was assessed by St. George's Respiratory Questionnaire (SGRQ) scale. Total score, ranged from 0 to 100, is the sum of points from all items. A higher value represents a worse outcome.
Change in lung imags of high resolution computed tomography (HRCT) from baseline | 24 weeks after treatment
  Lung images from HRCT will be analyzed to indicate the newly-derived pulmonary structure.
Acute exacerbation of idiopathic pulmonary fibrosis (IPF) | Within 24 weeks after treatment
  Frequency and severity of acute exacerbation of IPF will be evaluated.
Change in blood routine from baseline | Within 24 weeks after treatment.
  Number of cases or participants with abnormal laboratory test results will be evaluated.
Change in urine routine from baseline | Within 24 weeks after treatment.
  Number of cases or participants with abnormal laboratory test results will be evaluated.
Change in blood biochemistry from baseline | Within 24 weeks after treatment
  Number of cases or participants with abnormal laboratory test results will be evaluated.
Change in 12-lead Electrocardiogram (ECG) from baseline | Within 24 weeks after treatment
  Number of cases or participants with abnormal results wil be evaluated
Change in carcinoembryonic antigen (CEA) from baseline | 12 and 24 weeks after treatment
  CEA is a tumor marker used for early diagnosis of lung cancer.
Change in neuron-specific enolase (NSE) from baseline | 12 and 24 weeks after treatment
  NSE is a tumor marker significantly elevated in small cell lung cancer.
Change in cytokeratin-19-fragment (CYFRA21-1) from baseline | 12 and 24 weeks after treatment
  CYFRA21-1 is a tumor marker which has important value for the pathological classification and prognosis evaluation of lung cancer.
Change in squamous cell carcinoma antigen (SCC) from baseline | 12 and 24 weeks after treatment
  SCC is a specific marker for lung squamous cell carcinoma. Tumor markers are monitored to assess the safety.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No